CLINICAL TRIAL: NCT00320125
Title: Effects of Dairy Foods on Adolescent Pregnant Mothers and Their Newborns
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Dairy Council, Rosemont, Illinois, USA (Unknown)
Responsible Party: Gary M Chan, MD Primary Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 8818-01
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2008-10

CONDITIONS: Pregnancy
Keywords: Dairy; Calcium; Pregnancy; Fetus; Bone mineralization
MeSH Terms: interventions — Calcium; Dairy Products

ARMS (3):
- 1 (No Intervention): Usual diet
- 2 (Active Comparator): Orange juice fortified with calcium
  Interventions: Dietary Supplement: Orange juice plus calcium
- 3 (Active Comparator): Dairy products
  Interventions: Dietary Supplement: Dairy products

INTERVENTIONS:
Dietary Supplement: Orange juice plus calcium — > 1,200mg Ca (four glasses of orange juice plus calcium)per day
  Arms: 2
Dietary Supplement: Dairy products — > 1,200mg Ca (by consuming milk, yogurt, and cheese)
  Arms: 3

SUMMARY:
The purpose of the study is to evaluate the effects of different dietary calcium have on the pregnant teen mother and her newborn. We hypothesize that the higher calcium intake during pregnancy will result in higher bone mass in the newborn.

DETAILED DESCRIPTION:
Osteoporosis in the adult remains a significant public health problem. One of the major causes of osteoporosis is the inadequate calcium intake during the pediatric age range of birth to 20 years of age. We believe that this low calcium may start at birth since the fetus is actively accumulating calcium during the last trimester of pregnancy. Adolescents generally have poor calcium intake. Our study is to compare the newborn bone mass from adolescent mothers who are taking the recommended calcium intake from dairy foods or non-dairy foods such as orange juice during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant mothers aged 15 to 18 years, term gestation

Exclusion Criteria:

* Chronic disease such as hypertension, diabetes, medications that will affect calcium metabolism

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2002-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Newborn bone mass
Maternal dietary intakes

SECONDARY OUTCOMES:
Newborn body weight
Maternal blood pressure
Newborn blood for calcium, phosphate, vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Chan, MD, Principal Investigator — University of Utah
Locations (1):
- University Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Thomas M, Weisman SM. Calcium supplementation during pregnancy and lactation: effects on the mother and the fetus. Am J Obstet Gynecol. 2006 Apr;194(4):937-45. doi: 10.1016/j.ajog.2005.05.032. PMID 16580279
- [Result] Koo WW, Walters JC, Esterlitz J, Levine RJ, Bush AJ, Sibai B. Maternal calcium supplementation and fetal bone mineralization. Obstet Gynecol. 1999 Oct;94(4):577-82. doi: 10.1016/s0029-7844(99)00371-3. PMID 10511362
- [Result] Merrilees MJ, Smart EJ, Gilchrist NL, Frampton C, Turner JG, Hooke E, March RL, Maguire P. Effects of diary food supplements on bone mineral density in teenage girls. Eur J Nutr. 2000 Dec;39(6):256-62. doi: 10.1007/s003940070004. PMID 11395985
- [Result] Chan GM, McElligott K, McNaught T, Gill G. Effects of dietary calcium intervention on adolescent mothers and newborns: A randomized controlled trial. Obstet Gynecol. 2006 Sep;108(3 Pt 1):565-71. doi: 10.1097/01.AOG.0000231721.42823.9e. PMID 16946216
- [Derived] Kongwattanakul K, Duangkum C, Ngamjarus C, Lumbiganon P, Cuthbert A, Weeks J, Sothornwit J. Calcium supplementation (other than for preventing or treating hypertension) for improving pregnancy and infant outcomes. Cochrane Database Syst Rev. 2024 Nov 19;11(11):CD007079. doi: 10.1002/14651858.CD007079.pub4. PMID 39560075
- See also: national osteoporosis organization — http://www.nof.org
- See also: NIH osteoporosis resource center — http://www.osteo.org